CLINICAL TRIAL: NCT00714675
Title: Citrulline Supplementation in Elderly Malnourished and Hospitalised Subjects: Effects on Protein Metabolism
Brief Title: Citrulline and Protein Metabolism in the Malnourished Elderly People
Acronym: CIPROAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Kyowa Hakko Kogyo (Japan) providing the amino acids (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P070127
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Metabolism; Elderly
Keywords: citrulline; protein-energy malnutrition; aged; protein biosynthesis; amino acid
MeSH Terms: conditions — Protein-Energy Malnutrition | interventions — Citrulline; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Citrulline
  Interventions: Dietary Supplement: Citrulline
- 2 (Active Comparator): Amino acids
  Interventions: Dietary Supplement: Amino acids

INTERVENTIONS:
Dietary Supplement: Citrulline — 1 unit of 10 g L-Citrulline, 1 time on morning during 21 days
  Arms: 1
Dietary Supplement: Amino acids — 1 unit of an equivalent quantity of iso nitrogenous of non-essential amino acids(alanine, aspartate, glycine, serine, histidine, proline), 1 time on morning during 21 days.
  Arms: 2

SUMMARY:
The aim of this study is to evaluate the effects of a supplementation of citrulline for three weeks in elderly malnourished and hospitalised subjects on muscle protein synthesis.

DETAILED DESCRIPTION:
Malnutrition in the elderly causes an important public health problem because their response to re nutrition is highly decreased. Several experimental studies have shown that an amino acid named citrulline could avoid this, by restoring protein synthesis.

The treated group will receive each morning for three weeks a supplementation of 10 g of citrulline and the control group, non essential amino acids in iso-nitrogenous quantity to the 10g of citrulline.

During the three weeks of supplementation, clinical tolerance and physical exercise will be evaluated regularly.

On the 21st day, whole body protein synthesis rate in the post-absorptive state will be measured by the isotopic dilution of L-leucine (1-13C expressed in g / kg of lean mass / 24h) as well as other parameters of the protein turn-over in the post-absorptive and post-prandial state.

ELIGIBILITY:
Inclusion Criteria:

* elderly hospitalised in geriatric medicine or in following care and rehabilitation, moderately malnourished
* aged more than 70 years
* recent moderate undernutrition (30 g/l < albuminemia < 35 g/l and 18 < BMI < 22 or a score of the Mini Nutritional Assessment (MNA) < 17 with albuminemia > 30 g/l)
* ingesta of at least 20 kcal / kg / d and 0,8 g / kg / d of proteins

Exclusion Criteria:

* hospitalisation < 21d
* C reactive protein (CRP) > 50 mg / l
* end-stage cardiac insufficiency
* severe digestive incapacity
* renal insufficiency (Creatinine Clearance < 30 ml / mn)
* respiratory failure
* MMS < 18
* uncontrolled acute or chronic infectious pathology (HIV, tuberculosis)
* corticoids treatment
* evolutionary neoplasia
* palliative phase of severe pathology
* Mental Mini Score status of Folstein (MMS) < 8
* parenteral nutrition
* active chronic hepatitis or cirrhosis
* participation in another trial

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Whole body protein synthesis rate in the post-absorptive state measured by the isotopic dilution of L-leucine (1-13C expressed in g / kg of lean mass / 24h) | after 3 weeks of treatment

SECONDARY OUTCOMES:
clinical tolerance | Every day

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Melchior, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Emile Roux, Limeil-Brévannes, France

REFERENCES:
- [Background] Moinard C, Nicolis I, Neveux N, Darquy S, Benazeth S, Cynober L. Dose-ranging effects of citrulline administration on plasma amino acids and hormonal patterns in healthy subjects: the Citrudose pharmacokinetic study. Br J Nutr. 2008 Apr;99(4):855-62. doi: 10.1017/S0007114507841110. Epub 2007 Oct 22. PMID 17953788
- [Background] Osowska S, Duchemann T, Walrand S, Paillard A, Boirie Y, Cynober L, Moinard C. Citrulline modulates muscle protein metabolism in old malnourished rats. Am J Physiol Endocrinol Metab. 2006 Sep;291(3):E582-6. doi: 10.1152/ajpendo.00398.2005. Epub 2006 Apr 11. PMID 16608884